CLINICAL TRIAL: NCT06603649
Title: Evaluation of the Updated Procedure for the Management of Refractory Out-of-hospital Cardiac Arrests with SAMU 54 : the Revised ACEP Protocol in 02/2024
Brief Title: Evaluation of Updated Procedure for Management of Refractory Out-of-hospital Cardiac Arrests
Acronym: ACEP-V2
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, JAEGER Deborah, Principal investigator, Central Hospital, Nancy, France
Other Study IDs: 2024PI049
Record Dates: First submitted 2024-08-28; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Cardiac Arrest, Out-Of-Hospital
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: ECPR for out-of-hospital cardiac arrest — Patient with out-of-hospital cardiac arrest enrolled in the ECPR protocol

SUMMARY:
ECPR is a technique that has been rapidly developed in many cardiac arrest specialized centers In 2013, a specific management protocol was developed for patients in refractory out-of-hospital cardiac arrest around Nancy, France. To select patients with the best prognosis, the inclusion criteria defined were strict. This led to an over-selection of patients and a significant reduction in the number of eligible patients. A balance needed to be struck between over-selecting patients and maintaining the expertise of medical and paramedical teams in the field. In addition, it has also been shown that ECPR also increases the number of organs and transplants.

In February 2024, the criteria for inclusion in the protocol were redefined to include any witnessed non-traumatic cardiac arrest, whatever the initial rhythm. This simplification should enable more patients to be included in the procedure.

The aim of the study is to assess the patient's outcome

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital cardiac arrest
* enrolled in the ECPR program
* 18 years old or more
* Low-flow estimated <60minutes

Exclusion Criteria:

* traumatic cardiac arrest
* major comorbidities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting with refractory out-of-hospital cardiac arrest and enrolled in the ECPR program in Nancy, France.
  Inclusion criteria for the ECPR program are the following:
  * Age: 18-65 years
  * No major comorbidity
  * Witnessed non traumatic cardiac arrest
  * Low-flow to ECPR estimated of less than 60 minutes
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival | 90 days after cardiac arrest
  Survival rate of patients enrolled in the protocol

SECONDARY OUTCOMES:
Delays | From event to implementation of ECMO, in minutes, Up to 180 minutes
  Delay between cardiac arrest and ECPR implementation
Neurological outcome | 30 days and 90 days after cardiac arrest
  Evaluation of neurological outcome of survivors after cardiac arrest using the Rankin score

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided